CLINICAL TRIAL: NCT03982576
Title: Innovations to Prevent Relapse Among Low-income African American Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE5Y18
Record Dates: First submitted 2019-05-28; First posted 2019-06-11 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: 2-arm semi-pragmatic randomized design among recently quit smokers (N = 100). Random assignment (1:1 ratio, stratified by building and sex).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS Relapse Prevention (Experimental): Participants will receive 4 group sessions of a novel culturally specific, CBT-based intervention. They will also receive Path2Quit, a newly developed video-text program, which delivers 6 weeks of CS video messages (1-2 times/day) and provides 24/7 access to messages pulled from 3 keywords (HELP1, JONES, SLIP). Notably, CS relapse prevention will incorporate surface and deep structure elements,17 including race-matched interventionists, religion/spirituality, discussion of race-related stress, traditional values (e.g., collectivism), culturally specific recipes, etc.
  All participants will receive 4 weeks of nicotine replacement therapy (NRT; transdermal nicotine patches or nicotine gum).
  Interventions: Other: Nicotine replacement therapy (NRT); Behavioral: CS-CBT intervention; Behavioral: Path2Quit
- Standard Relapse Prevention (Active Comparator): Participants will receive 4 group sessions of a standard relapse prevention program, publicly available at smokefree.gov. Participants will also receive SmokefreeTXT, the NCI's 6-week fully automated text-based cessation program that is free to U.S. subscribers, and is available on smokefree.gov. Users can text one of 3 keywords (MOOD, CRAVE, or SLIP) to receive a relevant message from the system 24/7.
  All participants will receive 4 weeks of nicotine replacement therapy (NRT; transdermal nicotine patches or nicotine gum).
  Interventions: Other: Nicotine replacement therapy (NRT); Behavioral: Relapse prevention program; Behavioral: SmokefreeTXT

INTERVENTIONS:
Other: Nicotine replacement therapy (NRT) — 4 weeks of Transdermal nicotine patches or nicotine gum
Behavioral: CS-CBT intervention — 4 group sessions of a novel culturally specific, CBT-based intervention over 2 weeks
  Arms: CS Relapse Prevention
Behavioral: Path2Quit — Path2Quit is a newly developed video-text program, which delivers 6 weeks of CS video messages (1-2 times/day) and provides 24/7 access to messages pulled from 3 keywords (HELP1, JONES, SLIP).
  Arms: CS Relapse Prevention
Behavioral: Relapse prevention program — 4 group sessions of a standard relapse prevention program, publicly available at smokefree.gov
  Arms: Standard Relapse Prevention
Behavioral: SmokefreeTXT — NCI's 6-week fully automated text-based cessation program that is free to U.S. subscribers, and is available on smokefree.gov. Users can text one of 3 keywords (MOOD, CRAVE, or SLIP) to receive a relevant message from the system 24/7
  Arms: Standard Relapse Prevention

SUMMARY:
The purpose of this research is to study a relapse prevention program for adult former smokers in Northeast Ohio. The study will also look at how different people respond to the program. Participants asked to take part in this study because they contacted the team for help remaining tobacco-free or otherwise expressed interest in the program. The study includes completing surveys and receiving text messages to help stay tobacco free.

DETAILED DESCRIPTION:
The main objective of this study is to conduct a pilot study to assess the feasibility, acceptability, and initial efficacy/clinical significance of a tobacco relapse prevention intervention designed for low-income African Americans.

In this study, the team will estimate effect sizes for a culturally specific (CS) relapse prevention intervention compared to standard relapse prevention in a sample of low-income African American smokers and examine predictors of time to smoking relapse.

In a community-based clinical trial, adults who recently quit smoking (N=100) will be randomly assigned to one of two experimental conditions: (1) CS Relapse Prevention or (2) Standard Relapse Prevention. The primary outcome variables collected will include biochemically verified point prevalence abstinence (ppa) at 6-weeks and time to smoking relapse (TTR) over 3-months. This study will test daily hassles, cessation self-efficacy, coping strategies, and adherence to NRT as individual difference factors that may affect response to CS relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Adult smokers recruited from the community by study community navigator and flyers
* Self-identify as African American
* Report no tobacco smoking within the past 3-90 days and have a carbon monoxide (CO) reading of ≤ 3 ppm
* Have access to SMS texting
* Meet federal definitions of low-income

Exclusion Criteria:

- Study team will offer to enroll ineligible smokers in the publicly available smokefreeTXT (if applicable) or refer them to the Ohio state quitline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Biochemically verified point prevalence abstinence (ppa) | at 6-weeks from start of treatment
  Biochemically verified point prevalence abstinence (ppa) confirmed by breath carbon monoxide and saliva cotinine will confirm self-reported cessation at each follow-up.
Time to smoking relapse (TTR) | up to 3 months from start of treatment
  Time to smoking relapse (TTR) over a 3 month period

SECONDARY OUTCOMES:
Smoking urges | 20 minutes, 6-weeks follow-up, and 3-months from end of treatment.
  Measured through Weekly the Questionnaire of Smoking Urges (QSU) with scores ranging from 10-70, higher scores indicating greater urges.
Percent of participants adhering to nicotine replacement therapy (NRT) | 20 minutes, 6-weeks follow-up, and 3-months from end of treatment.
  Timeline follow-back (TLFB) instrument used to record daily use of NRT per day. The TLFB is a calendar that assesses daily smoking and NRT use. Based on participants' reconstruction of their smoking history, abstinence variables will be determined. For instance, if there has been no smoking in the 7 days preceding the assessment, the criterion for 7-day point prevalence abstinence (ppa) will be met.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Webb Hooper, PhD, Principal Investigator — Case Western Reserve University, Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Case Comprehensive Cancer Center, Cleveland, Ohio, United States